CLINICAL TRIAL: NCT02457052
Title: Impact of a Transportable Customizable and Scalable Sitting Positioning Device on Swallowing Disorders
Acronym: DATP-DEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 12 558 15; ID-RCB: 2013-A01351-44 (Registry Identifier: ANSM)
Record Dates: First submitted 2015-04-09; First posted 2015-05-29 (Estimated); Last update posted 2025-12-05 (Actual); Status verified 2019-07

CONDITIONS: Deglutition Disorders
Keywords: Medical device
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DATP + (Experimental): Introduction of a device allowing a custom sitting to help patients with swallowing disorders .
  Interventions: Device: DATP
- DATP - (No Intervention): No introduction of a device allowing a custom sitting to help patients with swallowing disorders .

INTERVENTIONS:
Device: DATP — Medical device allowing a custom sitting to help patients with swallowing disorders
  Arms: DATP +

SUMMARY:
When the seat is a vehicle for disabled person, postural adaptation methodology is known and, on prescription, there is possibility of financial support for technical posture assists. For people who use a standard seat, a chair for example, there is no satisfactory existing hardware.

A transportable customisable and scalable sitting positioning device (DATP device), to be placed on a standard seat, is a solution that might fit in the home, in specialized foster homes or in institutions for the elderly. Such a device has been developed but earnings on swallowing disorders have to be validated.

ELIGIBILITY:
Inclusion Criteria :

* Present a swallowing disorder authenticated by a score Dysphagia Handicap Index above 11
* Postural disorder authenticated by a score greater than 0 to at least 1 of the following 3 items to MCPAA: retroversion, obliquity and rotation of the pelvis
* Autonomy Conservation compatible with the use of different seats including standard seats
* Signing of informed consent

Exclusion Criteria:

* Postural disorder requiring the use of only one type of installation (wheelchair or hull)
* Spinal stiffness or non-reducible hips (spondylitis, osteosynthesis rod)
* Not included anthropometric dimensions between:

  * Basin with between 39 and 50 cm
  * femoral length between 42 and 52 cm
  * tibial length between 39 and 44 cm (46.5 with femoral recharge), measured with the shoes.
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-10; Primary Completion 2017-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in laryngeal movement during swallowing | One month
  Compare the laryngeal movement during swallowing in dysphagic population with DATP device compare to a population without device after one month of care.
  At Visit 1, patients were included and randomized
  1 month later the patients in both groups will be invited for specific education session positioning. The introduction of the device will be carried out before the meeting for patients DATP + group, which will include a training session in the use of DATP. Patients who have the DATP will be contacted by telephone within the first 15 days to verify compliance with the use of the device.
  All patients returned 1 month for the last visit.

SECONDARY OUTCOMES:
NIH Swallowing Safety Scale | One month
  The secondary outcomes are to evaluate the impact on other characteristics of swallowing, the posture, the acceptability of the device and the quality of life.
  Comparison before and after the treatment of dysphagia population with DATP compared to a population dysphagia.
Functional oral intake scale (FOIS) | One month
Adult sitting postural control measure (MCPAA) | One month
Quality questionnaire of patient's life | One month
  Using Short Form (36) Health Survey (SF-36)

CONTACTS AND LOCATIONS:
Overall Officials: Virginie WOISARD, MD; PHD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital, Toulouse, Toulouse, Midi-Pyrénées, France

REFERENCES:
- [Result] Woisard V, Costes M, Colineaux H, Lepage B. How a personalised transportable folding device for seating impacts dysphagia. Eur Arch Otorhinolaryngol. 2020 Jan;277(1):179-188. doi: 10.1007/s00405-019-05657-5. Epub 2019 Oct 4. PMID 31586257